CLINICAL TRIAL: NCT04874441
Title: Evaluation of the Effect of the Implementation of a Candida PCR Diagnosis Strategy on the Time Required to Obtain Results in Patients From Intensive Care Units With Suspected Systemic Invasive Candidiasis: Pilot Study
Brief Title: Candida PCR Diagnosis Strategy in Patients From Intensive Care Units
Acronym: CANDI-PCR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/19/0507
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Candida
Keywords: candidemia; Polymerase Chain Reaction; DNA; antifungal agents
MeSH Terms: conditions — Torulopsis; Candidemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blood culture-based diagnostic strategy (No Intervention): Patients from intensive care units with suspected invasive candidiasis initially treated with echinocandins and who benefited from a blood culture-based diagnostic strategy
- C. glabrata / krusei PCR diagnostic strategy (Experimental): Patients from intensive care units with suspected invasive candidiasis initially treated with echinocandins and who benefited from a diagnostic strategy based on C. glabrata / krusei PCR
  Interventions: Diagnostic Test: Diagnosis strategy based on C. glabrata / krusei PCR

INTERVENTIONS:
Diagnostic Test: Diagnosis strategy based on C. glabrata / krusei PCR — For diagnosis, a blood cultures and blood tubes for PCR will be collected and patients will be treated with echinocandins in the first instance with an early switch to fluconazole if the C. glabrata / krusei PCR is negative
  Arms: C. glabrata / krusei PCR diagnostic strategy

SUMMARY:
The aim of this study is to evaluate the implementation of a new technique for invasive candidiasis diagnosis by PCR. The main objective will be to evaluate the effect of this strategy on the time required to obtain results in patients from intensive care units with suspected systemic invasive candidiasis. This PCR method could allow an antifungal switch to be made earlier, limiting the appearance of resistance and reducing the cost of antifungals for healthcare facilities.

DETAILED DESCRIPTION:
Invasive candidiasis is a serious infection caused by yeasts of the genus Candida sp. Their incidence is increasing, particularly in intensive care. The prognosis is severe and depends on the early initiation of adequate antifungal treatment. At present, the diagnosis of invasive candidiasis is difficult since blood culture, the reference technique, has major limitations due to its low sensitivity, as well as very long delays in obtaining results. As a consequence, suspected invasive candidiasis is often treated empirically with echinocandins, resulting in the development of resistance and extremely high costs for health care facilities. The switch to treatments such as fluconazole is often delayed, although this molecule is effective on most Candida species except C. krusei and glabrata and is much less expensive than echinocandins.

For these reasons, the present study developed faster and more efficient methods to diagnose Candida krusei and glabrata species, based on the detection of DNA in the blood by PCR, allowing an earlier switch from echinocandins to Fluconazole.

The patients included will be divided into 2 groups: one group of patients will benefit from a diagnostic strategy based on blood culture (reference technique for the detection of Candida) and another group of patients will benefit from a diagnostic strategy based on this new PCR technique. The main objective will be to evaluate the effect of the PCR strategy on the time to obtain results and on the switch of antifungal agents. After inclusion, patients will be followed up at day 14, day 28 until discharge (or 3 months if the patient is still hospitalised).

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated or benefiting from a social protection system
* Patient (or his/her trusted person) having given free and informed written consent to the investigating physician
* Non-neutropenic patient hospitalised in the Toulouse University Hospital intensive care unit.
* Patient with suspected invasive candidiasis for whom a blood culture for fungal infection diagnosis was taken and for whom an empirical treatment with echinocandin at an adapted dose was implemented.

Exclusion Criteria:

* Patients under guardianship or trusteeship, persons under court protection
* Pregnant or breastfeeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Reporting delay | 14 days after blood sample taken
  the time (in hours) required for the results to be returned in relation to the time of sample collection

SECONDARY OUTCOMES:
mortality at Day 28 | 28 days after blood sample taken
  Mortality rates will be taken 28 days after taking blood samples for Candida diagnosis in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Pamela CHAUVIN, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Uh Toulouse, Toulouse, Occitanie, France